CLINICAL TRIAL: NCT05039541
Title: Feasibility Study: Using the Alio Medical REmoteMOnitoring System (RMS) to Non-InvasivelyMonitor Subjects With EnD-Stage REnaL DiseaseSubjects
Brief Title: The ReModel IHC Study for ESRD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GW-12
Record Dates: First submitted 2021-08-18; First posted 2021-09-09 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Dialysis Access Malfunction
Keywords: vascular access monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ESRD Patients (Experimental): ESDR Patients will wear the Alio Device over their vascular access for either I) the duration of their dialysis session in clinic or II) for a 90 day period.
  Interventions: Device: Alio Device

INTERVENTIONS:
Device: Alio Device — Subjects will wear the Alio device over their vasculature.

SUMMARY:
There will be two phases of this study. The phases of this study may occur simultaneously. In Phase I, eligible subjects will be asked to acutely wear the Alio Medical RMS SmartPatch during regularly scheduled dialysis sessions. Subjects will have a pre- and post-dialysis blood draw(s), vitals collected, and monitoring throughout the dialysis sessions. The SmartPatch will be removed from the location(s) where it is placed following the post-dialysis blood draw.

In Phase II, subjects will be asked to wear a SmartPatch for up to 90 days. Subjects will be trained on the use of the Alio Medical RMS and be provided a system for them to utilize at home. Patches will be changed at a minimum of once every 7 days.

DETAILED DESCRIPTION:
There will be two phases of this study. The phases of this study may occur simultaneously. For Phase I subjects' consent will be completed via RedCap in person upon their first study related dialysis visit. In Phase I, eligible subjects will be asked to acutely wear the Alio Medical RMS SmartPatch during regularly scheduled dialysis sessions.The SmartPatch automatically records data and uploads it to the Alio Cloud. Subjects will have a pre- and post-dialysis blood draw(s), vitals collected, and monitoring throughout the dialysis sessions. The SmartPatch will be removed from the location(s) where it is placed following the post-dialysis blood draw.

For Phase II consent will be completed via RedCap either in clinic during a visit to pick up supplies or via email and digital communication if the subject is unable to drive to the clinic location. In Phase II, subjects will be asked to wear a SmartPatch for up to 90 days. The exact wear time will be documented on the case report form (CRF). Any request for specific wear times and frequency of SmartPatch changes will be documented prior to study start on the consent form or CRF. This will be done to enable continuous non-invasive measurements of the patient metrics (e.g., hemoglobin (Hb), hematocrit (Hct),heart rate (HR), and other relevant dialysis labs or vitals). Subjects will be trained on the use of the Alio Medical RMS and be provided a system for them to utilize at home. Patches will be changed at a minimum of once every 7 days.

In addition to At-Home device use, subjects will also be participating in acute data collection during one (or more) of their in-clinic or at home dialysis sessions. Approximately every two to four weeks over the course of Phase 2, subjects will have a pre- and post-dialysis blood draw(s), vitals collected, and SmartPatch monitoring.

Further, any procedures, hospitalizations or additional relevant labs/imaging will also be collected for the purposes of comparing the Alio Medical RMS to standard of care assessments. At the end of the study, subjects maybe asked to complete a short survey on their experience with the Alio Medical RMS. Select study staff will have access to Alio Medical RMS study data for the purposes of comparing this information to the clinical standard(s) collected.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80.
* Maintenance dialysis for ESRD for at least 6 months.
* Dialysis via an AVF or AVG in an arm location.
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.
* Can speak, read and communicate in English.
* Willing and able to wear the SmartPatch as instructed and comply with the visits, tests, and schedule of evaluations.

Exclusion Criteria:

* Hospital admission within last 30 days which, in the opinion of the physician or study staff, could potentially affect the subject's ability to participate in the study procedures.
* Pseudoaneurysm on the measured AV access.
* Liver disease associated with serum albumin levels less than 35 g/L.
* History of acute illness episode that, in the opinion of their physician or study staff, could potentially affect study data being collected.
* Significant fluid overload (patient > 3kg above dialysis dry weight at start of dialysis session)
* Subjects with novel materials for their AVF or hAVG, such as HeRO grafts, chest-wall AVFs
* Subjects with rapid-use grafts (e.g., AVflo™ or Gore® Acuseal)
* Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study if, in the judgement of the study staff, participation in this study could potentially affect the quality of study data.
* Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.
* The Study Doctor(s) determine(s) that the subject is not eligible for participation in this research study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Alio device comparison to Hct via blood draws | through study completion, an average of 1 year
  Compare the Alio device to dialysis clinic blood lab values drawn before and after dialysis. The Hematocrit value collected will be compared to the Alio device.
Alio device comparison to K+ via blood draws | through study completion, an average of 1 year
  Compare the Alio device to dialysis clinic blood lab values drawn before and after dialysis. The Potassium value collected will be compared to the Alio device.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kraus, MD, Principal Investigator — Intermountain Health Care
Locations (1):
- Intermountain Dialysis, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No